CLINICAL TRIAL: NCT04340583
Title: Subjective Sleep Quality and Prevalence of Sleep Disorders in Patients With Severe Asthma
Brief Title: Subjective Sleep Quality and Sleep Disorders in Patients With Severe Asthma
Status: Terminated | Type: Observational
Why Stopped: organization problems
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2289 CE
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-01

CONDITIONS: Asthma
Keywords: Sleep disorder; Monoclonal therapy; Anxiety; Depression
MeSH Terms: conditions — Asthma; Sleep Wake Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchial asthma is characterized by the presence of symptoms that vary over time and of severity. Asthma symptoms tend to worsen at night and in the early hours of the morning, and the presence of nocturnal symptoms is an important indicator of therapeutic intervention in order to control the severity of the disease. Aim of the study is to investigate sleep disorders and quality, as well as and depressive and anxiety symptoms in patients affected by severe asthma before and after 6 months of treatment with monoclonal therapy. An observational, cohort, prospective, monocentric study will be conducted to evaluate subjective quality of sleep at baseline and post monoclonal treatment.

DETAILED DESCRIPTION:
Rationale

Bronchial asthma is a heterogeneous and highly prevalent disease; moreover, it represents one of the main cost of the Italian National Health Care System. According to international guidelines, asthma is characterized by the presence of symptoms such as wheezing, dyspnoea, chest tightness and / or cough, and limitation of expiratory air flow, that vary over time and of severity.

The main therapy consists of the use of inhaled corticosteroids in order to reduce airway inflammation; however, in conditions characterized by frequent exacerbations, patients take oral corticosteroids (OCS) cyclically or chronically to control their symptoms. Asthma symptoms tend to worsen at night and in the early hours of the morning, and the presence of nocturnal symptoms is an important indicator of therapeutic intervention in order to control the severity of the disease.

Several studies have shown that nocturnal symptoms, such as cough and dyspnoea, are associated with circadian oscillations of airway inflammation and physiological variables, with consequent air flow limitation of and bronchial hyperreactivity. Moreover, it is known that patients receiving OCS are subjected to significant alterations of the hypothalamic-pituitary-adrenergic axis function, therefore the assumption of these drugs could cause a modification of the circadian rhythm.

Since sleep fragmentation that accompanies the worsening of nocturnal asthmatic symptoms is probably caused by the degree of severity of nocturnal bronchoconstriction, it is possible that severe asthmatic patients have greater bronchoconstriction and therefore more disturbed sleep.

Subjects with severe asthma, the 5-10% of the total asthmatic population, report symptoms that persist despite inhalation therapy, and have many exacerbations, Emergency Room access or hospitalizations.

These patients use systemic steroids at least twice a year due to asthmatic exacerbations and / or continuous therapy with systemic steroids for at least 6 consecutive months, with the development of side effects such as high blood pressure, overweight, meta-steroid diabetes and osteoporosis.

In the last ten years, the availability of alternative therapies such as monoclonal antibodies, which block the inflammatory cascade at different levels (Anti Immunoglobulin E, Anti interleukin-5 (II-5)e anti receptor Il-5) has allowed to reduce the dosage of steroid therapy up to its complete suspension.

Obstructive Sleep Apnoea (OSA) is one of the most common asthma comorbidities, especially severe, affecting about 26% of patients. When evaluated with polysomnography, the prevalence of OSA is equal to 88% in patients with severe asthma and 58% in those with moderate asthma.

It seems that OSA could contribute to asthma exacerbations, to diurnal and nocturnal symptoms and to the scarce quality of life; it also seems to modulate airway inflammation and remodeling. Asthmatic patients with OSA show a greater decline in Forced Expiratory Volume in the first second (FEV1) over time than non-OSA, and Continuous Positive Airways Pressure (CPAP) treatment seems to slow down this deterioration. Serrano Pariente et al. have demonstrated that 6 months CPAP treatment improves the outcomes of Asthma in patients with moderate OSA. Finally, a recent study has shown that patients with poorly controlled asthma tend to have worse sleep quality and greater diurnal sleepiness. The same study has demonstrated a higher prevalence of depressive symptoms in female patients with poorly controlled asthma.

Aim of the study is to investigate sleep disorders and quality, as well as and depressive and anxiety symptoms in patients affected by severe asthma before and after 6 months of treatment with monoclonal therapy.

Primary outcome is to evaluate subjective quality of sleep at baseline and post treatment.

Secondary outcomes are: to verify pre and post treatment: the presence of insomnia, respiratory disorders, circadian rhythm disorders, diurnal sleepiness or anxiety and depression symptoms.

Inclusion criteria:

* Diagnosis of severe persistent asthma
* Systemic steroids treatment for at least 6 months and/or ≥2 exacerbations in the last year
* Need to initiate monoclonal antibody therapy according to guidelines
* Age ≥18 years
* Signed Informed consent
* Patients able to collaborate in the required procedures

Exclusion criteria:

Diagnosis of cognitive impairment Study Design An observational, cohort, prospective, monocentric study will be conducted. Patients will be enrolled c/o the Pneumology Division of the Clinical and Scientific Institute Maugeri of Tradate.

Data will be collected at baseline (T0) and after 6 months of therapy with one monoclonal antibody (omalizumab, mepolizumab or benralizumab) (T6).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe persistent asthma
* Systemic steroids treatment for at least 6 months and/or ≥2 exacerbations in the last year
* Need to initiate monoclonal antibody therapy according to guidelines
* Age ≥18 years
* Signed Informed consent
* Patients able to collaborate in the required procedures

Exclusion Criteria:

* Diagnosis of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referral to medical clinic
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
subjective quality of sleep | 6 months
  Pittsburgh Sleep Quality Index score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

SECONDARY OUTCOMES:
Insomnia | 6 months
  Insomnia Severity Index score ranging from 0 to 28 where lower scores denote no problems
respiratory disorders | 6 months
  Berlin questionnaire High Risk: if there are 2 or more categories where the score is positive, Neck circumference, Obesity, Snoring, Age, Sex (Nosa) Questionnaire,The score ranges from 0 to 17 and the patient has a high probability of OSA if they have a NoSAS score of 8 or higher
circadian rhythm disorders | 6 months
  Morningness-Eveningness Questionnaire Scores can range from 16-86. Scores of 41 and below indicate "evening types". Scores of 59 and above indicate "morning types". Scores between 42 and 58 indicate "intermediate types
diurnal sleepiness | 6 months
  Epworth Sleepiness Scalerange ranging from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life
anxiety | 6 months
  State Trait Anxiety Inventory ranging from 20 to 80, with higher scores correlating with greater anxiety.
depression | 6 months
  Beck Depression Inventory ranging from 0 to 63 were higher scores indicate more severe depressive symptoms.
sleep quality | 6 months
  Maugeri Sleep Quality and Distress Inventory ranging from 17 to 51 were higher scores indicate the presence of greater sleep-related distress.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Study Chair — Istituti Clinici Maugeri
Locations (1):
- Istituti Clinici Maugeri Pneumologia, Tradate, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collomp R, Labsy Z, Zorgati H, Prieur F, Cottin F, Do MC, Gagey O, Lasne F, Collomp K. Therapeutic glucocorticoid administration alters the diurnal pattern of dehydroepiandrosterone. Endocrine. 2014 Aug;46(3):668-71. doi: 10.1007/s12020-013-0122-9. Epub 2013 Dec 18. PMID 24347241
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Campos FL, de Bruin PFC, Pinto TF, da Silva FGC, Pereira EDB, de Bruin VMS. Depressive symptoms, quality of sleep, and disease control in women with asthma. Sleep Breath. 2017 May;21(2):361-367. doi: 10.1007/s11325-016-1422-0. Epub 2016 Oct 29. PMID 27796717